CLINICAL TRIAL: NCT07111039
Title: Pilot Study to Compare Airway Pressure Release Ventilation (APRV) to Conventional Mechanical Ventilation (CMV) During Anesthesia for Robotic-Assisted Gynecological and Genitourinary Operative Procedures
Brief Title: Compare Airway Pressure Release Ventilation (APRV) to Conventional Mechanical Ventila
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays impactful to study operations
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23490
Record Dates: First submitted 2025-07-02; First posted 2025-08-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Gynecologic Cancer; Genitourinary Cancer
MeSH Terms: conditions — Urogenital Neoplasms | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- APRV compared to CMV (Experimental): APRV will be tested during anesthesia in 12 patients undergoing robotic-assisted gynecological or genitourinary surgical procedures for definitive cancer treatment, who will also receive CMV.
  Interventions: Other: Airway Pressure Release Ventilation; Other: Conventional Mechanical Ventilation

INTERVENTIONS:
Other: Airway Pressure Release Ventilation — APRV
Other: Conventional Mechanical Ventilation — CMV

SUMMARY:
This is a pilot study to determine if pulmonary function (lung compliance and ventilation/perfusion matching) is improved using APRV during general anesthesia, compared to the standard CMV. APRV will be tested during anesthesia in 12 patients undergoing robotic-assisted gynecological or genitourinary surgical procedures for definitive cancer treatment, who will also receive CMV.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed gynecological or genitourinary cancer.
* Subjects will have the physiologic reserve to undergo a robotic-assisted gynecological or genitourinary surgical procedure that uses anesthesia via Airway Pressure Release Ventilation and via Conventional Mechanical Ventilation.
* Adults (≥18 years old)
* ECOG performance status ≤ 2.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Vulnerable subjects will not be enrolled for this study.
* Patients who have COPD and are on oxygen at home or who have COPD requiring routine daily inhalers or daytime oxygen are excluded.
* Patients who have history of major lung resection are excluded.
* Patients with body mass index (BMI) >50 are excluded.
* Patients with pulmonary infection within the past 2 months of screening are excluded.
* The availability of oxygen to a fetus during this experimental procedure has not been established. Therefore, patients known to be pregnant per operating room (OR) policy will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Optimal intra-operative ventilatory settings - Inspiratory Pressure | At surgery
  Determination of the optimal intra-operative ventilatory settings for inspiratory pressure, expiratory pressure, inspiratory-expiratory time ratio and inspired oxygen concentration, that result in the best possible measured pulmonary function (i.e., compliance and gas exchange).
Optimal intra-operative ventilatory settings - Expiratory Pressure | At surgery
  Determination of the optimal intra-operative ventilatory settings for inspiratory pressure, expiratory pressure, inspiratory-expiratory time ratio and inspired oxygen concentration, that result in the best possible measured pulmonary function (i.e., compliance and gas exchange).
Optimal intra-operative ventilatory settings - Inspiratory-expiratory time ratio | At surgery
  Determination of the optimal intra-operative ventilatory settings for inspiratory pressure, expiratory pressure, inspiratory-expiratory time ratio and inspired oxygen concentration, that result in the best possible measured pulmonary function (i.e., compliance and gas exchange).
Optimal intra-operative ventilatory settings - Inspired oxygen concentration | At surgery
  Determination of the optimal intra-operative ventilatory settings for inspiratory pressure, expiratory pressure, inspiratory-expiratory time ratio and inspired oxygen concentration, that result in the best possible measured pulmonary function (i.e., compliance and gas exchange).

CONTACTS AND LOCATIONS:
Overall Officials: David Thrush, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States